CLINICAL TRIAL: NCT03237962
Title: Effectiveness of High Flow Nasal Nannula on Exercise Endurance Among Patients During Pulmonary Rehabilitation
Brief Title: High Flow Nasal Cannula During Pulmonary Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Hui-Ling Lin, Assistant Proffesor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NMRPD1F0731
Record Dates: First submitted 2017-07-16; First posted 2017-08-03 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: High flow nasal cannula; Pulmonary rehab; Pulmonary rehabilitation; Nasal cannula; Exercise endurance; Oxygen Therapy; COPD; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Cannula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Flow Nasal Cannula (Experimental): Patients are randomly assigned into High flow nasal cannula group for the exercise training
  Interventions: Device: High Flow Nasal Cannula
- Nasal Cannula (Experimental): Patients are randomly assigned into nasal cannula group for the exercise training.
  Interventions: Device: Nasal Cannula

INTERVENTIONS:
Device: High Flow Nasal Cannula — High Flow Nasal Cannula (HFNC) is an oxygen device that increases oxygenation and washes out CO2 within the dead space, it was also clinically used to correct hypoxemia, hypercapnia and respiratory failure.By providing flow rate that is similar to or higher than the patient's inspiratory flow, HFNC is able to provide ventilatory support. To produce stable oxygen concentration, HFNC entrains less air in order to reach the preset value.
  Other Names: HFNC
  Arms: High Flow Nasal Cannula
Device: Nasal Cannula — Nasal cannula is an oxygen therapy device that has been commonly used as treatment for patients with hypoxemia. With the adjustable flow of 1-6Lpm, the concentration of the oxygen differs as the breathing pattern of the patient changes.
  Arms: Nasal Cannula

SUMMARY:
The primary purpose of this study is to compare and assess the immediate and long-term effects on pulmonary rehabilitation training with the usage of HFNC or conventional oxygen therapy device.

The hypotheses was, with high flow nasal cannula usage while exercising, the physiological outcome measurements would be better than conventional oxygen therapy device. Also, the usage of HFNC can immediately increase patient's exercising endurance and decrease dyspnea caused by exercising.

DETAILED DESCRIPTION:
Pulmonary Rehabilitation is one of the most recommended methods to improve the muscle function of COPD patients. By exercise training, even patients with severe COPD can increase muscle strength, improve skeletal muscle function and enhance exercise endurance. Due to improvements in exercise endurance, when exercising at a higher intensity, ventilation support and dynamic hyperinflation would slightly decrease which leads to less dyspnea during exercise. Continuously exercising can also increase the motivation to exercise, reduce mood irritability and psychological burden caused by symptoms. By exercising, patient's health status can be both improved physically and mentally.

High Flow Nasal Cannula (HFNC) is a non-invasive ventilatory device that provides stable oxygen concentration, temperature (37℃) and humidity (Relative Humidity: 100%). Humidity provided by the HFNC reduces irritation caused by the high flow, which leads to the increase of user's tolerance with the device. With the half-closed system formed by a nasal prong, when the high flow enters the upper airway, continue positive airway pressure would be formed.

Subjects enrolled into this study are required to join a 6-week pulmonary rehabilitation program. Before starting the program, subjects were randomly assigned to high flow nasal cannula group and conventional oxygen therapy group. When exercising, the nasal cannula group would receive an oxygen flow of 3 - 5L to maintain SpO2>90% and the HFNC group with high flow setting of 45-50Lpm along with oxygen flow of 3-5L also to maintain SpO2>90%. When joining the pulmonary rehabilitation program, patients are required to exercise for approximately 45 minutes per session. When exercising, changes in the degree of dyspnea, quadriceps blood flow and hemodynamics are assessed. After 6-week of the exercise training, all the parameters will again be assessed and compared to the primary data that was collected from the beginning of the program.

ELIGIBILITY:
Inclusion Criteria:

* Age > 55 years
* COPD patients with confirmed pulmonary function test results of FEV1<70%
* Regular follow-up at the pulmonary medicine clinic
* Stable condition without acute exacerbation
* No pulmonary rehabilitation training within a year
* None oxygen usage at home
* No smoking history or quit smoking
* Inform consent signed

Exclusion Criteria:

* Fever (Body Temperature >37.5°C)
* Acute infection symptoms
* Unstable cardiovascular status (Eg: Blood pressure >150/100 mmHg after medication usage, angina pectoris, or abnormal ECG)
* Activity restrictions due to orthopedic or neuromuscular disease

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Cardiac Output in L/min | Changes from baseline to 6 weeks and 12 weeks
  Heart rate and stroke volume will be combined to report cardiac output in L/min

SECONDARY OUTCOMES:
COPD Assessment Test (CAT) | Changes from baseline to 6 weeks and 12 weeks
  Questionnaire designed to evaluate COPD patient's quality of life.
Modified Medical Research Council (mMRC) Dyspnea Scale | Changes from baseline to 6 weeks and 12 weeks
  Scale to determine the breathlessness of COPD patients during their daily activity
The maximum inspiratory pressure in cmH2O | Changes from baseline to 6 weeks and 12 weeks
  The maximum inspiratory pressure in cmH2O represents the strength of the abdominal and expiratory muscles
The maximum expiratory pressure in cmH2O | Changes from baseline to 6 weeks and 12 weeks
  The maximum expiratory pressure in cmH2O
Tissue Saturation Index | Changes from baseline to 6 weeks and 12 weeks
  Tissue Saturation Index measured by near-Infrared spectroscopy
Total Hemoglobin | Changes from baseline to 6 weeks and 12 weeks
  Total Hemoglobin measured by near-Infrared spectroscopy
Borg Scale | Changes from baseline to 6 weeks and 12 weeks
  Scale examining the level of dyspnea or the shortness of breath during exercise

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Ling Lin, MSc, Principal Investigator — Chang Gung University
Locations (2):
- Taiwan (2):
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
  - Chang Gung Memorial Hospital, Taoyuan District